CLINICAL TRIAL: NCT01754688
Title: Determining Prevalence of Acute Bilirubin Encephalopathy in Developing Countries
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1109M04335
Record Dates: First submitted 2012-06-21; First posted 2012-12-21 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Hyperbilirubinemic Encephalopathy
Keywords: Acute Bilirubin Encephalopathy; Bilirubin Induced Neurologic Dysfunction score; Hearing Test; Neonate
MeSH Terms: conditions — Kernicterus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Jaundice infants: Bilirubin Induced Neurologic Dysfunction II score

SUMMARY:
The investigators hypothesize that a new BIND (Bilirubin Induced Neurologic Dysfunction) scoring method adapted for the developing world (BIND II, developed by our team for use by health care workers), with additional modifications for community use (the community BIND, C-BIND), will improve the ability to identify infants with ABE and to distinguish ABE from other common causes of neonatal morbidity and mortality compared to currently available survey tools.

DETAILED DESCRIPTION:
This is a minimal risk observational cross sectional study to validate a scoring tool, the BIND II, to diagnose ABE. Babies with suspected jaundice (n=709) and without jaundice (n=125) will be enrolled. Data from a hearing test, physical exam, and laboratory tests will be used to compare with the results from the scoring tool.

The BIND II will be done by the physician examining the infant before the ABR study is done as it is simply a scored physical exam focused on signs of acute bilirubin encephalopathy. The BIND II will be done by the physician examining the patient at/near the time of the ABR testing. The physician will be a consultant when possible but when not possible it will be another trained physician and that will be documented.

The BIND II will be done by the physician trained by a pediatric consultant or Drs. Slusher/Olunsanya. The ABR will be performed by audiology technicians under the direction of Dr. Olunsanya. Since Dr. Olunsanya will see some of the infants during this time and, therefore, not be blinded to their clinical status, Dr. Steve Shapiro, a pediatric neurologist with expertise in reading ABE in infants and children with ABE/Kernicterus, will read all ABR while remaining blinded to clinical details of each infant.

The mothers will then be interviewed by trained community workers during either a follow-up visit at the hospital or at a later time during the admission if the baby is still admitted. The mothers will be shown photographs, video, and will listen to audio recordings as part of the interview process. These images and recordings are used to ask questions about the mother's perception of her baby's condition at the time of the initial admission. The community workers will complete the Community- or C-BIND form and determine a rating. This rating will then be compared with the physicians' BIND II score. The community worker will be blinded to the results of the BIND II and the ABR reading.

Community health worker will be defined as a lay person not formally trained as a registered nurse or doctor but may have training as an assistant nurse although this will not be required. Lay workers qualified to be community health workers but not yet working as community health workers will be able to participate as community health workers in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible to participate in the study if all of the following conditions exist:

  1. At time of birth, neonates who are ≥ 35 weeks gestational age or

     ≥ 2250 grams if gestational age unavailable.
  2. ≤ 14 days old
  3. Parent or guardian has given consent for the infant to participate

Exclusion Criteria:

1. Infants with a condition requiring urgent referral to another facility for treatment not available at the hospital study site.
2. Infants being admitted for a surgical procedure only without an underlying medical illness.
3. Infants who have a condition that requires no blood draws for treatment of their problem and only reason for blood draw would be study enrollment. -

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates admitted to Massey Street Children's Hospital
Sampling Method: Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2012-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Slusher, MD, Study Chair — University of Minnesota
Locations (1):
- Massey Street Children's Hospital, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out at Massey Street Children's Hospital and the surrounding community in Lagos, Nigeria. Recruitment began in January 2013 and ended in March 2015.
Groups:
- Neonates: observational cross sectional study to validate a scoring tool, the BIND II, to diagnose ABE
Period: Overall Study
Arm/Group | Neonates
Started | 624
Completed | 624
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neonates
Number analyzed (Participants) | 624
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Estimated Gestational Age (weeks)
  weeks | 39 [38 to 40]
Sex/Gender, Customized [Number; unit: participant]
  Male | 416
  Female | 202
  Unknown | 6
Admission Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 3.0 [2.6 to 3.3]

OUTCOME MEASURES:

1. Primary Outcome: Bilirubin Induced Neurologic Dysfunction II Score (BIND II)
Description: The original BIND was developed in the USA to score infants with Acute Bilirubin Encephalopathy using a focused physical exam (primarily neurologic) and history to determine the degree of encephalopathy a infant with jaundice displayed. The BIND has been adapted for Low-Middle-Income Countries.
  The bilirubin-induced neurologic dysfunction (BIND) scoring algorithm was developed, assigning 0, 1, 2 or 3 points to each of the four sections to indicate none, mild, moderate, or severe abnormalities in an infant's mental status, muscle tone, cry, and eye/facial findings. Each of the four sections has a maximum score of 3, giving a total BIND score range of 0 to 12. Higher scores indicate worsening signs of acute neurotoxicity associated with excessive hyperbilirubinemia.
Time Frame: Birth to 14 days
Population: observational cross sectional study to validate a scoring tool, the BIND II, to diagnose ABE
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Neonates
Number analyzed (Participants) | 584
units on a scale | 1 [0 to 4]

2. Secondary Outcome: Community Bilirubin Induced Neurologic Dysfunction Score (C-BIND)
Description: We will translate the BIND II into lay language and have community workers administer it using pictures and/or short videos along with simple questions to the same infants that the doctors performed the BIND II, and compare the score of the community workers with those of the physicians to validate this score. The community workers will not examine the infants. They will do everything through questions and pictures and/or videos.
  The bilirubin-induced neurologic dysfunction (BIND) scoring algorithm was developed, assigning 0, 1, 2 or 3 points to each of the four sections to indicate none, mild, moderate, or severe abnormalities in an infant's mental status, muscle tone, cry, and eye/facial findings. Each of the four sections has a maximum score of 3, giving a total BIND score range of 0 to 12. Higher scores indicate worsening signs of acute neurotoxicity associated with excessive hyperbilirubinemia.
Time Frame: Birth to 14 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Neonates
Number analyzed (Participants) | 624
units on a scale | 3 [1 to 4]

ADVERSE EVENTS:
Arm/Group | Neonates
Serious Adverse Events (participants affected / at risk) | 0/624
Other Adverse Events (participants affected / at risk) | 0/624

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No